CLINICAL TRIAL: NCT02226939
Title: A Randomised, Double-blind, Placebo Controlled Trial With 200 mg BILN 2061 ZW Given p.o. at Two Consecutive Days Bid to Investigate the Antiviral Efficacy, Pharmacokinetics, Safety in Patients With Cirrhosis and Chronic Hepatitis C
Brief Title: Antiviral Efficacy, Pharmacokinetics and Safety of BILN 2061 ZW in Patients With Cirrhosis and Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 605.9
Record Dates: First submitted 2014-08-26; First posted 2014-08-27 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Liver Cirrhosis; Hepatitis C, Chronic
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis C, Chronic | interventions — BILN 2061

ARMS (2):
- BILN 2061 ZW (Experimental)
  Interventions: Drug: BILN 2061 ZW
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BILN 2061 ZW
  Arms: BILN 2061 ZW
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to assess the antiviral efficacy, pharmacokinetics, and tolerability of 200 mg BILN 2061 ZW in a polyethylene glycol 400 (PEG 400: ethanol) drinking solution given orally for two days bid to patients with cirrhosis and chronic Hepatitis C Virus (HCV) infection

ELIGIBILITY:
Inclusion Criteria:

* Female or male sex, age of 18 years or older
* Chronic Hepatitis C virus (HCV) infection
* Liver biopsy consistent with active HCV infection obtained within the last 36 months.
* No previous clinical evidence of decompensated cirrhosis. Present cirrhosis status consistent with grade A, according to Child-Turcotte-Pugh classification, confirmed at screening
* No evidence of significant gastroesophageal varices (> grade 1 or other risk factors) according to fiberoptic endoscopy performed within the last 12 months
* No evidence of Hepatocellular carcinoma (HCC) by ultrasound performed at screening
* Written informed consent consistent with International Committee on Harmonization (ICH) / Good Clinical Practice (GCP) and local legislation given prior to any study procedures
* HCV of genotype I
* HCV load greater than 50,000 copies messenger ribonucleic acid (mRNA) per ml serum at screening

Exclusion Criteria:

* Women of childbearing potential or breastfeeding women. Postmenopausal women less than 6 months after last menses, surgically sterilized or hysterectomised less than 3 months after operation or not having negative serum pregnancy test
* Males not using an adequate form of contraception (condom, sterilization at least 6 months post operation) in case their partner is of childbearing potential (criteria see above) and is not using an adequate form of contraception (hormonal contraceptives, oral or injectable/ implantable, intra-uterine device (IUD))
* Any other or additional plausible cause for chronic liver disease, including the presence of other viruses known or suspected to cause hepatitis
* Evidence of gastroesophageal varices
* Any histological evidence of hepatocytic dysplasia
* Following serological constellations: Hepatitis B surface (HBs)-Ag positive OR anti-Hepatitis B core (HBc) positive with anti- HBs negative OR anti-HAV IgM positive OR anti-Human immunodeficiency Virus (HIV) positive
* History of abuse of alcohol within the past twelve months
* Planned or concurrent usage of any other pharmacological therapy at screening, including any antiviral therapy
* Any concurrent infectious disease requiring antimicrobial treatment
* History of malignancy (except for previously cured squamous cell or basal cell carcinoma of the skin)
* Usage of any investigational drug within thirty (30) days prior to enrolment; or the planned usage of an investigational drug during the course of the current study
* Known hypersensitivity to drugs
* Inability to comply with the protocol
* Prior or present Child´s B or C liver diseases -

  * Bilirubin - refer to following exclusion criterion
  * Prothrombin time < 70%
  * Albumin < 3.5 g/dl
  * Clinical evidence of ascites
  * Clinical evidence of encephalopathy
* Clinically apparent jaundice or a total bilirubin or alkaline phosphatase exceeding 2.0 x upper limit of normal (ULN) at screening
* ALT or AST >= 10 x ULN at screening
* A platelet count of less than 80.000 platelets per mm3 at screening
* White blood cell count of less than 2,000 cells per mm3 at screening
* AFP > 100 ng/ml
* Splenectomy
* Positive test for illicit or unprescribed drugs or medications at screening. Positive test for cannabis may be allowed if the investigator assesses this result not as clinically significant
* Patients with any clinically significant laboratory abnormalities based on the investigator's medical assessment at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2002-09; Primary Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Virus load (VL) as determined by number of copies of HCV mRNA per ml serum | up to day 14
  Cobas Amplicor HCV Monitor v 2.0 (HCM-2.0, Roche Diagnostics)

SECONDARY OUTCOMES:
Number of patients with relevant drug-induced changes in alanine aminotransferase (ALT) | up to day 14
Number of patients with relevant drug-induced changes in aspartate aminotransferase (AST) | up to day 14
Number of patients with relevant drug-induced changes in vital signs (pulse rate, systolic and diastolic blood pressure) | up to day 14
Number of patients with relevant drug-induced changes in electrocardiography (ECG) | up to day 14
Number of patients with relevant drug-induced changes in routine laboratory tests | up to day 14
Number of patients with adverse events | up to 35 days
Maximum concentration in plasma after a single dose administration (Cmax) | up to day 4
Area under the plasma concentration-time curve from t = 0 to t = .τ rate (AUC0-τ) | up to day 4
Time to reach Cmax following a single dose administration (tmax) | up to day 4
Total oral clearance of drug from plasma after oral administration, divided by F (CL/F) | up to day 4
Apparent volume of distribution during the terminal elimination phase (Vz/F) | up to day 4
Assessment of tolerability by investigator on a 4-point scale | day 3